CLINICAL TRIAL: NCT06305936
Title: The Feasibility and Acceptability of a Plant-Based Diet in People With Rheumatoid Arthritis - A Randomized Feasibility Study
Brief Title: Feasibility Study: Plant Based Diet to Patients With Rheumatoid Arthritis
Acronym: PLATE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Collaborators: Glostrup University Hospital, Copenhagen (Other)
Responsible Party: Principal Investigator, Allan Linneberg, Director, Professor, MD, PhD, Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: PLATE H-23042292
Record Dates: First submitted 2024-02-27; First posted 2024-03-12 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Rheumatoid Arthritis
Keywords: feasibility study; rheumatoid arthritis; plant-based food diet intervention
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Methods; Diet, Plant-Based

STUDY DESIGN:
Intervention Model Description: Randomised feasibility study of an intervention group, receiving 100% plant-based diet and a control group
Who Masked: Investigator, Outcomes Assessor
Masking Description: Not possible to blind participants and study staff delivering the intervention to allocation status, whereas all outcome data is planned to be collected by blinded outcome assessors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): As part of the 4-week intervention in the feasibility study, the intervention group will receive 1) Educational materials (videos) 2) Participation in a cooking workshop with introduction to PBD meals, including recipes, and 3) Daily delivered PBD dinner meal during the four weeks.
  Interventions: Other: Intervention with 100% plant-based diet
- Control group (No Intervention): The control group will be asked to maintain habitual diet and lifestyle. In addition, they will follow the same outcome assessments as the intervention group.

INTERVENTIONS:
Other: Intervention with 100% plant-based diet — The intervention consists of three key components: 1) Educational materials (videos), 2) Participation in a cooking workshop introducing plant-based meals, complete with recipes, and 3) Daily delivery of plant-based dinner meals over a four-week period. The remaining meals during the period are modified by the participant to also adhere to a 100% plant-based composition.
  Other Names: Diet intervention
  Arms: Intervention group

SUMMARY:
In this feasibility study, our primary goal is to assess the practicality of implementing a plant-based food diet intervention for individuals with rheumatoid arthritis (RA). The intervention consists of three key components: 1) Educational materials (videos), 2) Participation in a cooking workshop introducing plant-based meals, complete with recipes, and 3) Daily delivery of plant-based dinner meals over a four-week period. This comprehensive investigation covers the testing of recruitment procedures, randomization, intervention elements, outcome assessments, and participant retention.

Adopting a daily plant-based diet involves introducing several new plant-based foods and making adjustments to the existing diets of patients with RA. Consequently, the feasibility study will also aim to explore the acceptability of the intervention and whether a full-scale RCT is practically possible.

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is a common chronic autoimmune disease requiring lifelong pharmacological treatment and causing significant burden to the patient and society. Evidence has suggested that it is important that patients take an active role in their self-management to improve their overall health and quality of life. Effective self-management strategies often involve changes in lifestyle. We have previously conducted a lifestyle intervention study to reduce sedentary behavior and increase physical activity in 150 patients with RA. An individually tailored intervention motivating patients to self-manage their arthritis by reducing sedentary behavior and replacing it with light-intensity physical activity reduced disease activity, e.g., levels of pain and fatigue. Nutrition may be another important part of self-management strategies in patients with RA. Emerging evidence suggests that an anti-inflammatory diet may reduce disease activity and improve quality of life among patients with RA.3 Compared to a diet including animal foods, a Plant-Based Diet (PBD) is believed to include less of the pro-inflammatory, and more of the anti-inflammatory, ingredients, and thus may have the potential to reduce disease activity in patients with RA.

Our overall and long-term aim is to test and evaluate the effect of a PBD intervention on disease activity in patients with RA in a later randomized controlled trial (RCT). As a first step towards this, we wish to investigate strengths and limitations of the planned intervention, which introduces a PBD to patients with RA.

Thus, in a feasibility study, we aim to investigate the feasibility of the intervention, including recruitment procedures, randomization, intervention elements, outcome assessments and retention. Following a daily PBD will involve inclusion of several new plant-based foods and changes in earlier diets for patients with RA. As such, the feasibility study will also aim to investigate acceptability of the intervention, including how people with RA respond to the intervention elements and how a PBD affect their daily lives (e.g. how easy is it to prepare plant-based foods, how desirable is it to eat, and how does it affect digestion). Ultimately, the findings from this feasibility study will provide crucial insights into whether a full-scale randomized controlled trial (RCT), designed to evaluate the effects of a 100% plant-based diet on patients with RA, is a feasible and realistic undertaking.

ELIGIBILITY:
Inclusion Criteria:

* Disease Activity Score with 28 Joint Counts (DAS28) between 2.0-3.2
* A rheumatoid arthritis diagnosis of minimum 1 year
* Under stable pharmaceutical treatment for at least 4 months and with no planned change in treatment within 8 weeks

Exclusion Criteria:

* Daily smokers
* Diabetes Mellitus
* Pregnancy / planned pregnancy
* Lactation
* Prednisolone treatment
* DAS28 below 2.0 and above 3.2
* Current dietary habits resembling intervention diet (e.g., 100% plant based diets)
* Participation in other intervention studies or clinical trials via the rheumatology outpatient clinic that will affect their adherence to plant based diets
* Not able to eat ad libitum meals because of e.g., allergy
* Unable to understand the informed consent and study procedures
* Alcohol and/or drug abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-02-15 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Feasibility and Intervention Fidelity in Implementing a Plant-Based Food Diet Intervention - Evaluating the feasibilty of included objectively measured outcomes and self-administered questionnaires | 3 months
  This study aims to evaluate the feasibility of implementing a plant-based food diet (PBD) intervention by assessing participant acceptability and feasibility in achieving desired outcomes. Feasibility testing will involve specific objective outcome assessments, including both objectively measured outcomes and self-administered questionnaires outlined below as secondary outcomes.
Evaluation of Study Acceptance | 3 months
  This study assesses the acceptability of the study protocol from qualitative methods through focus group interviews, exploring topics such as the effectiveness of food delivery methods and participants' perceptions of the plant-based diet intervention.
Recruitment | 3 months
  Recruitment rates will be calculated as the proportion of patients randomised/proportion of patients eligible
Retention | 3 months
  Retention rates will be calculated as the proportion of patients providing the outcomes of interest/proportion of patients randomised
Intervention adherence | 3 months
  Adherence of intervention protocol will be calculated as the number of received optional elements of the intervention out of the total number of optional intervention elements available

SECONDARY OUTCOMES:
Disease Activity Score (DAS28) | 3 months
  Estimate of Disease Activity Score (mean and SD) in patients with rheumatoid arthritis. The Disease Activity Score 28 (DAS28) is a composite index used in rheumatology to assess disease activity in patients with rheumatoid arthritis. The DAS28 is a quantification of tender and swollen joints within the hands, shoulders, elbows, wrists, and knees. These assessments, in conjunction with CRP values obtained from blood samples and the self-reported global Visual Analog Scale (VAS) score, will be incorporated into the computation of DAS28. The DAS28 ranges from 0 to 10, with higher scores indicating higher disease activity.
Fatigue: Bristol Rheumatoid Arthritis Fatigue (BRAF MDQ) | 3 months
  Assessed in each participant at baseline and follow-up. The BRAF MDQ covers several domains fatigue, including living, cognitive, emotional and physical fatigue. 20 items are included in the questionnaire, where you can obtain a total fatigue score.
Pain (VAS) | 3 months
  Assessed in each participant at baseline and follow-up. Participants' pain levels will be measured by the Visual Analogue Scale (VAS), which transforms the subjective experience of pain to a measurable quantity.
Sleep | 3 months
  Assessed in each participant at baseline and follow-up. The Pittsburgh Sleep Quality Index (PSQI) is a self-rated questionnaire that assesses sleep quality and disturbances. The time interval is 1 month interval. Nineteen individual items generate a component score (subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction). The sum of these generates one global score.
Anxiety/depression | 3 months
  Assessed in each participant at baseline and follow-up. The Hospital Anxiety and Depression Scale (HADS) is used to screen for psychological distress in medical outpatients through self-report. It is a 14-item self-report scale that measures the presence of symptoms related to both anxiety (7 items) and depression (7 items) during the past week.
Physical function | 3 months
  Assessed in each participant at baseline and follow-up. The Multidimensional Health Assessment Questionnaire (MD-HAQ) is applied to measure self-reported functional status over the previous seven days on ten items covering dressing, rising, eating, walking, hygiene, reach, grip and everyday activities.
Impact of rheumatoid arthritis (RA) | 3 months
  Assessed in each participant at baseline and follow-up. The Rheumatoid Arthritis Impact of Disease (RAID) score is a valid tool used to measure the impact of RA in different domains. The domains include pain, function, fatigue, sleep, disturbance, emotional and physical wellbeing.
The EuroQuality of Life (EQ-5D) | 3 months
  Assessed in each participant at baseline and follow-up. The EuroQuality of Life (EQ-5D) generic health index will be used as a health index to calculate the health profile. It questionnaire comprises a five-part questionnaire and a visual analogue self-rating scale.
Height | 3 months
  Assessed in each participant at baseline and follow-up to calculate BMI.(Unit: CM)
Weight | 3 months
  Assessed in each participant at baseline and follow-up to calculate BMI. (Unit: Kg)
Waist- and hip circumference | 3 months
  Assessed in each participant at baseline and follow-up to calculate waist-hip ratio
Disease activity | 3 months
  Assessed in each participant at baseline and follow-up. Assessing joint inflammation and damage in patients with rheumatoid arthritis (RA) using ultrasound imaging from ultrasound examinations. These are performed to gain an additional objectively view on the disease activity. This is performed on wrist, metacarpophalangeal joint (MCP) 1-5, proximal interphalangeal joint (PIP) 1-5, ankle joint and metatarsophalangeal joint (MTP) 2-5. The joints will be scored from 0-3 after the Ultrasound Scoring System for Rheumatoid Arthritis by the Outcome Measures in Rheumatology (OMERACT). Assessed in each participant at baseline and follow-up.
Body composition | 3 months
  Assessed in each participant at baseline and follow-up. Anthropometry reflected by body fat percentage (%) assessed by bioimpedance (unit is estimated per cent fat mass).
Quantification of tender and swollen joints | 3 months
  Assessed in each participant at baseline and follow-up. A quantification of tender and swollen joints within the hands, shoulders, elbows, wrists, and knees will be undertaken by a designated project nurse. Applied for the compution of DAS28.
C-reactive Protein (CRP) | 3 months
  Assessed in each participant at baseline and follow-up. Blood samples will be drawn by a project nurse to get a picture of current health status at baseline and end of study. (Unit: mg/L)
Hemoglobin | 3 months
  Assessed in each participant at baseline and follow-up. Blood samples will be drawn by a project nurse to get a picture of current health status at baseline and end of study. (Unit: mmol/L)
Leukocytes | 3 months
  Assessed in each participant at baseline and follow-up. Blood samples will be drawn by a project nurse to get a picture of current health status at baseline and end of study. (Unit: mia/L)
Thrombocytes | 3 months
  Assessed in each participant at baseline and follow-up. Assessed in each participant at baseline and follow-up. Blood samples will be drawn by a project nurse to get a picture of current health status at baseline and end of study. (Unit: mia/L)
Hemoglobin (HbA1c) | 3 months
  Assessed in each participant at baseline and follow-up. Blood samples will be drawn by a project nurse to get a picture of current health status at baseline and end of study. (Unit: mmol/mol)
D-vitamin | 3 months
  Assessed in each participant at baseline and follow-up. Blood samples will be drawn by a project nurse to get a picture of current health status at baseline and end of study. (Unit: nmol/L)
Low-density lipoprotein (LDL) | 3 months
  Assessed in each participant at baseline and follow-up. Blood samples will be drawn by a project nurse to get a picture of current health status at baseline and end of study. (Unit: mmol/L)
High-density lipoprotein (HDL) | 3 months
  Assessed in each participant at baseline and follow-up. Blood samples will be drawn by a project nurse to get a picture of current health status at baseline and end of study. (Unit: mmol/L)
Triglyceride | 3 months
  Assessed in each participant at baseline and follow-up. Blood samples will be drawn by a project nurse to get a picture of current health status at baseline and end of study. (Unit: mmol/L)
Total cholesterol | 3 months
  Assessed in each participant at baseline and follow-up. Blood samples will be drawn by a project nurse to get a picture of current health status at baseline and end of study. (Unit: mmol/L)

CONTACTS AND LOCATIONS:
Overall Officials: Allan Linneberg, Ph.D., Principal Investigator — Bispebjerg Hospital
Locations (2):
- Denmark (2):
  - Center for Clinical Research and Prevention, BispebjergH, Frederiksberg
  - The Department of Rheumatology and Spine Diseases, Copenhagen Center for Arthritis Research (COPECARE), Rigshospitalet, Glostrup, Glostrup Municipality

IPD SHARING:
Plan to Share IPD: No